CLINICAL TRIAL: NCT06918743
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase II Clinical Study Evaluating the Efficacy and Safety of RSS0393 Ointment Local Administration in Adults With Chronic Plaque Psoriasis
Brief Title: To Evaluate the Efficacy and Safety of RSS0393 Ointment in Patients With Plaque Psoriasis Phase II Study
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RSS0393Oint-201
Record Dates: First submitted 2025-03-24; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-02

CONDITIONS: Psoriatic Subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment group 1 (Experimental): RSS0393 ointment 0.01%
  Interventions: Drug: RSS0393 ointment
- Treatment group 2 (Experimental): RSS0393 ointment 0.03%
  Interventions: Drug: RSS0393 ointment
- Treatment group 3 (Placebo Comparator): RSS0393 ointment placebo
  Interventions: Drug: RSS0393 ointment placebo

INTERVENTIONS:
Drug: RSS0393 ointment — RSS0393 ointment 0.01%
  Arms: Treatment group 1
Drug: RSS0393 ointment — RSS0393 ointment 0.03%
  Arms: Treatment group 2
Drug: RSS0393 ointment placebo — RSS0393 ointment placebo
  Arms: Treatment group 3

SUMMARY:
To evaluate the efficacy and safety of RSS0393 ointment in patients with plaque psoriasis Phase II study

ELIGIBILITY:
Inclusion Criteria:

1. The age of signing the informed consent must be ≥18 years old and ≤75 years old, male or female
2. At screening, body mass index [BMI= weight (kg)/height 2 (m2)]≥18.0kg/m2
3. A history of plaque psoriasis ≥6 months prior to randomization
4. At screening and baseline, the BSA of the affected area was 2%-20% (including both ends), PASI score ≥2, PGA score ≥2.
5. The subject voluntarily signs informed consent before the start of any procedures related to the study, is able to communicate with the investigator smoothly, understands and is willing to complete the study in strict compliance with the requirements of the clinical study protocol;
6. A fertile female subject or a male subject whose partner is a fertile woman who has not had a child, plans to donate sperm/eggs from the date of signing the informed consent to 8 weeks after the last dose, and voluntarily uses highly effective contraceptive methods

Exclusion Criteria:

1. Present with any of the following medical history or concomitant diseases:

   1. Diagnosis of other types of psoriasis other than plaque psoriasis during subject screening, Such as guttate psoriasis, pustular psoriasis, erythrodermic psoriasis, articular psoriasis, or drug-induced psoriasis
   2. the subject has other skin diseases or conditions that the investigator determines may affect the evaluation of the relevant endpoint of this study
   3. any other persistent active autoimmune disease, Including but not limited to rheumatoid arthritis, systemic lupus erythematosus, scleroderma or polymyositis, multiple sclerosis or other central demyelinating diseases, primary Sjogren's syndrome, immune deficiency syndromes (such as Felty's syndrome);
2. There are the following important medical history or underlying diseases that affect safe

   1. The subject has a history of any active malignancy or malignancy in the 5 years prior to the screening visit, except skin squamous cell carcinoma or basal cell carcinoma or cervical cancer in situ that has been cured after treatment;
   2. Participants with a history of depression and/or who were clinically deemed to be at risk of suicide during the screening and baseline periods;
   3. Active infection within 2 weeks prior to baseline requiring systemic anti-infective therapy, or severe infection or systemic infection within 4 weeks prior to baseline requiring intravenous anti-infective therapy or hospitalization due to infection, or other chronic, recurrent, or active infections deemed by the investigator not suitable for participation in the study;
   4. had any surgery within 1 month prior to screening, or had not recovered as determined by the investigator, or planned any surgery during the study period;
   5. Currently has an active tuberculosis infection, or chest radiography indicates the presence of an active tuberculosis infection;
   6. any serious, progressive, uncontrolled cardiovascular or cerebrovascular, respiratory, liver, kidney, gastrointestinal, blood, neurological, or psychiatric disorders, or medical measures, medical conditions, etc. that may affect study participation, or may place subjects at undue risk, as determined by the investigator;
3. At the time of screening, laboratory tests and/or 12-lead electrocardiogram showed the following:

   1. Hemoglobin < 100.0 g/L (male) or < 90.0 g/L (female);
   2. White blood cell count < 3.0×109/L;
   3. Neutrophil count < 1.5×109/L;
   4. Platelet count < 100×109/L;
   5. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2.5 times the upper limit of normal (ULN);
   6. Total bilirubin (TBIL) > 1.5 times the upper limit of normal (ULN); g) The estimated glomerular filtration rate (eGFR) calculated by the simplified MDRD formula (see Appendix 13.5 for details) is < 60 mL/min/1.73 m², or the serum creatinine is outside the normal range, and the investigator determines that participation in this study is not appropriate;
   7. Hepatitis B surface antigen (HBsAg), human immunodeficiency virus antibody (HIV), syphilis antibody test, anti-hepatitis C virus (HCV) antibody test positive; If HBsAg is negative but hepatitis B core antibody (HBcAb) positive and hepatitis B virus deoxyribonucleic acid (HBV DNA) positive or above the upper limit of normal;
   8. 12-lead electrocardiogram examination indicates clinically significant abnormalities that may affect the safety of the subject, including but not limited to acute myocardial ischemia, myocardial infarction, severe arrhythmia, or significant QTc prolongation (QTc>500 ms).
4. General situation

   1. Pregnant or lactating women, defined as the female state from pregnancy to termination of pregnancy and positive blood test for human chorionic gonadotropin (β-HCG) during the screening period;
   2. Allergic to the investigational drug or any ingredient in the investigational drug
   3. a history of alcohol or illicit drug abuse in the year prior to screening
   4. received a live attenuated vaccine in the 12 weeks prior to randomization, intended to receive a live attenuated vaccine during the study period, or participated in a vaccine clinical trial in the 12 weeks prior to randomization
   5. Donate approximately 500 mL blood within 8 weeks prior to randomization or have a blood donation plan during the study period
   6. Subjects who are expected to have excessive exposure to natural/artificial light, sunbathing, or other light emitting diodes (leds) in the treatment area during treatment in this study; The investigators determined that there were conditions that affected the safety and efficacy evaluation of the study drugs or other conditions that were not suitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with a clinician's overall assessment (PGA) response (defined as a PGA score of 0 (clear) or 1 (nearly clear) with ≥2 points improvement from baseline) | 8weeks

SECONDARY OUTCOMES:
Proportion of participants who achieved at least 75% improvement (PASI 75) from baseline; | 14weeks
The proportion of subjects with PGA response at each visit | 14weeks
Absolute and percentage changes in PASI scores at each visit compared to baseline; | 14weeks
The proportion of subjects who achieved PGA 0 or 1 score at each visit | 14weeks
The time of the subject reached PASI 50 within 12 weeks | 14weeks
The proportion of participants who achieved at least a 50% improvement (PASI 50) in PASI scores from baseline at each visit | 14weeks
Percentage of participants who achieved at least a 90% improvement (PASI 90) from baseline in PASI scores at each visit | 14weeks
Absolute and percentage changes in the most intense itch digital score (WI-NRS) from baseline at each visit ; | 14weeks
The proportion of subjects with baseline involvement in the intererase area and intererase PGA (I-PGA) score ≥2 who achieved an I-PGA response (defined as an I-PGA of 0 or 1 with ≥2 points improvement from baseline) at each visit | 14weeks
The proportion of subjects with baseline involvement and I-PGA score ≥2 who achieved I-PGA score 0 at each visit | 14weeks
Absolute value of change in skin quality of life index (DLQI) from baseline at each visit | 14weeks

IPD SHARING:
Plan to Share IPD: Undecided